CLINICAL TRIAL: NCT02413398
Title: A Multicenter, Double-Blind, Placebo-Controlled, Parallel Group, Randomized, Phase III Study to Evaluate the Glycemic Efficacy and Renal Safety of Dapagliflozin in Patients With Type 2 Diabetes Mellitus and Moderate Renal Impairment (CKD 3A) Who Have Inadequate Glycemic Control.
Brief Title: A Study to Evaluate the Effect of Dapagliflozin on Blood Glucose Level and Renal Safety in Patients With Type 2 Diabetes
Acronym: DERIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1690C00024
Record Dates: First submitted 2015-04-07; First posted 2015-04-09 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental): 10 mg Tablets, Oral, Once daily, 24 weeks
  Interventions: Drug: Dapagliflozin 10 mg
- Placebo (Placebo Comparator): Matching placebo to Dapagliflozin 10 mg tablet. Oral, Once daily, 24 weeks
  Interventions: Drug: Matching Placebo for Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Tablets administered orally once daily for 24 weeks. Randomization will be stratified by pre-enrolment anti-hyperglycemic therapy
  Other Names: Farxiga™
  Arms: Dapagliflozin
Drug: Matching Placebo for Dapagliflozin — Matching Placebo for Dapagliflozin tablets administered orally once daily for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this clinical research study is to determine whether dapagliflozin can improve (decrease) blood glucose values in patients with Type 2 diabetes and moderate renal impairment.This study will be conducted at approximately 100 centres from countries across North America and European regions. It is planned to randomize a total of 302 patients.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged ≥18 years and <75 years.
* History of T2DM for more than 12 months.
* Inadequate glycemic control, defined as HbA1c ≥7.0% and ≤11%
* Stable anti-diabetic treatment regimen
* Renal impairment: CKD 3A

Exclusion Criteria:

* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period.
* History of diabetic ketoacidosis or hyperosmolar nonketotic coma.
* Severe uncontrolled hypertension defined as SBP ≥180 mmHg and/or Diastolic Blood Pressure (DBP) ≥110 mmHg
* Any of the following Cardiovascular (CV)/Vascular Diseases within 3 months of prior to signing the consent at visit 1:

Myocardial infarction, Cardiac surgery or revascularization(CABG/PTCA), Unstable angina, Unstable heart failure (HF), HF New York Heart Association (NYHA) Class IV,Transient ischemic attack (TIA) or significant cerebrovascular disease, Unstable or previously undiagnosed arrhythmia.

* History of any biopsy or imaging verifying intercurrent kidney disease (such as glomerular nephritis or sign of renal artery stenosis) other than diabetic nephropathy or diabetic nephropathy with nephrosclerosis.
* Significant hepatic disease, including, but not limited to, chronic active hepatitis and/or severe hepatic insufficiency.
* Ongoing treatment with any SGLT2-inhibitor, GLP-1 analogue, or rapid/short acting insulins at screening.
* Participation in another clinical study with an Investigational Product (IP) during the last 30 days prior to signing the consent at visit 1.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (80):
- United States (25):
  - Research Site, Huntsville, Alabama
  - Research Site, Burbank, California
  - Research Site, Chula Vista, California
  - Research Site, Concord, California
  - Research Site, Fullerton, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Gatos, California
  - Research Site, Newport Beach, California
  - Research Site, Salinas, California
  - Research Site, Miami, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Brownsburg, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Monroe, Louisiana
  - Research Site, Flint, Michigan
  - Research Site, Jackson, Michigan
  - Research Site, Chesterfield, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Manassas, Virginia
- Bulgaria (6):
  - Research Site, Blagoevgrad
  - Research Site, Botevgrad
  - Research Site, Kozloduy
  - Research Site, Kyustendil
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (16):
  - Research Site, Red Deer, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Concord, Ontario
  - Research Site, Courtice, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, London, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Czechia (7):
  - Research Site, Cheb
  - Research Site, Hořovice
  - Research Site, Krnov
  - Research Site, Kutná Hora
  - Research Site, Ostrava
  - Research Site, Prague
  - Research Site, Praha Klanovice
- Italy (8):
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Chieti Scalo
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, San Giovanni Rotondo
- Poland (7):
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Mrągowo
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Tczew
  - Research Site, Wroclaw
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Ferrol
  - Research Site, La Laguna (Tenerife)
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pozuelo de Alarcón
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Fioretto P, Del Prato S, Buse JB, Goldenberg R, Giorgino F, Reyner D, Langkilde AM, Sjostrom CD, Sartipy P; DERIVE Study Investigators. Efficacy and safety of dapagliflozin in patients with type 2 diabetes and moderate renal impairment (chronic kidney disease stage 3A): The DERIVE Study. Diabetes Obes Metab. 2018 Nov;20(11):2532-2540. doi: 10.1111/dom.13413. Epub 2018 Jul 10. PMID 29888547
- See also: Redacted Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3689&filename=D1690C00024-Clinical%20Study%20Protocol-v%204.0_redacted_final_1.pdf
- See also: Redacted SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3689&filename=D1690C00024-Statistical-Analysis-Plan-Edition-2_redacted_final_PDF_A.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin 10mg QD: 10 mg Tablets, Oral, Once daily, 24 weeks
- Placebo QD: Matching Placebo, 10 mg Tablets, Oral, Once daily, 24 weeks
Period: Overall Study
Arm/Group | Dapagliflozin 10mg QD | Placebo QD
Started | 160 | 161
Completed | 156 | 154
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other Eligibility criteria | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matching Placebo, 10 mg Tablets, Oral, Once daily, 24 weeks
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10mg QD | Placebo | Total
Number analyzed (Participants) | 160 | 161 | 321
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (6.22) | 66.2 (6.49) | 65.8 (6.36)
Age, Customized [Count of Participants; unit: Participants]
  < 65 Years | 64 | 46 | 110
  >= 65 Years | 96 | 115 | 211
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 139
  Male | 91 | 91 | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 2 | 0 | 2
  Asian | 5 | 8 | 13
  Black Or African American | 11 | 12 | 23
  Other | 1 | 1 | 2
  White | 141 | 140 | 281
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.6 (4.7) | 31.6 (5.0) | 32.1 (4.9)
Estimated Glomular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 51.8 (4.1) | 51.6 (3.8) | 51.7 (3.9)
Urine Albumin-to-Creatinine Ratio (UACR) [Mean (Standard Deviation); unit: mg/g] — Population: 159/160 subjects in the Dapaglifozin group had an enrolment UACR value.
  mg/g
    number analyzed (Participants) | 159 | 161 | 320
    (all) | 226.91 (566.67) | 246.52 (775.49) | 236.78 (678.81)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24
Description: To compare the mean change from baseline in HbA1c between dapagliflozin 10 mg and placebo, after 24 weeks of oral administration of double-blind treatment in patients with type 2 diabetes, CKD stage 3A, and moderate renal impairment (CKD 3A; eGFR 45-59 mL/min/1.73m^2). The "number analyzed" (142 dapaglifozin, 134 placebo) represents the number with change from baseline available at Week 24.
Time Frame: Baseline, Week 24
Population: For glycaemic measurements (HbA1c and FPG), all measurements after the first dose of rescue medication were excluded. For other non-glycaemic measurements (body weight and SBP), all measurements after the first dose of rescue medication were included.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 142 | 134
percent | -0.37 (0.10) | -0.03 (0.10)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Difference in adjusted mean change from baseline (MMRM model); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.53 to -0.15], Standard Error of Mean 0.10

2. Secondary Outcome: Adjusted Mean Percent Change From Baseline in Total Body Weight at Week 24.
Description: To compare the mean percent change from baseline in total body weight between dapagliflozin 10 mg and placebo, after 24 weeks of oral administration of double-blind treatment in patients with type 2 diabetes, CKD stage 3A, and moderate renal impairment (CKD 3A; eGFR 45-59 mL/min/1.73m^2). The "number analyzed" represents the number with change from baseline available at Week 24.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 149 | 146
percent change | -3.42 (0.32) | -2.02 (0.32)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Difference in adjusted mean percent change from baseline (MMRM); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.43, 95% CI 2-sided [-2.15 to -0.69], Standard Error of Mean 0.37

3. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24.
Description: To compare the mean change from baseline in FPG between dapagliflozin 10 mg and placebo, after 24 weeks of oral administration of double-blind treatment in patients with type 2 diabetes, CKD stage 3A, and moderate renal impairment (CKD 3A; eGFR 45-59 mL/min/1.73m^2). The "number analyzed" represents the number with change from baseline available at Week 24.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 135 | 134
mg/dL | -21.46 (5.20) | -4.87 (5.13)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Difference in adjusted mean change from baseline versus placebo (MMRM); Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -16.59, 95% CI 2-sided [-26.73 to -6.45], Standard Error of Mean 5.15

4. Secondary Outcome: Adjusted Mean Change From Baseline in Seated Systolic Blood Pressure (SBP) at Week 24.
Description: To compare the mean change from baseline in seated systolic blood pressure (SBP) between dapagliflozin 10 mg and placebo, after 24 weeks of oral administration of double-blind treatment in patients with type 2 diabetes, CKD stage 3A, and moderate renal impairment (CKD 3A; eGFR 45-59 mL/min/1.73m^2). The "number analyzed" represents the number with change from baseline available at Week 24.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 146 | 145
mmHg | -4.8 (1.5) | -1.7 (1.5)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Difference in adjusted mean change from baseline vs. placebo (MMRM); Test type: Superiority; p < 0.050, Mixed Models Analysis; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-6.3 to 0.0], Standard Error of Mean 1.6

ADVERSE EVENTS:
Time Frame: Non-serious AEs were included up to the last day of double-blind treatment + 4 days. SAEs were recorded from the time of Informed Consent through included up to the last day of double-blind treatment + 30 days (or to the end of the 3-week follow-up period, whichever came first).
Arm/Group | Dapagliflozin 10mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/161
Serious Adverse Events (participants affected / at risk) | 9/160 | 14/161
Other Adverse Events (participants affected / at risk) | 0/160 | 0/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg QD (N=160) | Placebo (N=161)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (2)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT02413398/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT02413398/SAP_001.pdf